CLINICAL TRIAL: NCT00686075
Title: A Phase 1/2a, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, Immunogenicity and Vaccine-like Viral Shedding of MEDI-534, a Live, Attenuated Intranasal Vaccine Against Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV3), in Healthy 6 to < 24 Month-old Children and in 2 Month-old Infants
Brief Title: A Study to Evaluate the Safety, Tolerability, Immunogenicity and Vaccine-like Viral Shedding of MEDI-534, Against Respiratory Syncytial Virus (RSV) and Parainfluenza Virus Type 3 (PIV3), in Healthy 6 to <24 Month-old Children and in 2 Month-old Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP178
Record Dates: First submitted 2008-05-23; First posted 2008-05-29 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Respiratory Syncytial Virus (RSV); Parainfluenza Virus Type 3 (PIV3); MEDI-534

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- MEDI-534, Cohort 1 (Experimental): Participants aged 6 to less than (<) 24 months will receive MEDI-534, 10^5 median tissue culture infectious dose (TCID50) by intranasal route at Month 0, 2, and 4.
  Interventions: Biological: MEDI-534, Cohort 1
- Placebo, Cohort 1 (Placebo Comparator): Participants aged 6 to <24 months will receive placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Other: Placebo, Cohort 1
- MEDI-534, Cohort 2 (Experimental): Participants aged 6 to <24 months will receive MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Biological: MEDI-534, Cohort 2
- Placebo, Cohort 2 (Placebo Comparator): Participants aged 6 to <24 months will receive placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Other: Placebo, Cohort 2
- MEDI-534, Cohort 3 (Experimental): Participants aged 2 months will receive MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Biological: MEDI-534, Cohort 3
- Placebo, Cohort 3 (Placebo Comparator): Participants aged 2 months will receive placebo matched to MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Other: Placebo, Cohort 3
- MEDI-534, Cohort 4 (Experimental): Participants aged 2 months will receive MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Biological: MEDI-534, Cohort 4
- Placebo, Cohort 4 (Placebo Comparator): Participants aged 2 months will receive placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Other: Placebo, Cohort 4
- MEDI-534, Cohort 5 (Experimental): Participants aged 2 months will receive MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Biological: MEDI-534, Cohort 5
- Placebo, Cohort 5 (Placebo Comparator): Participants aged 2 months will receive placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Interventions: Other: Placebo, Cohort 5

INTERVENTIONS:
Biological: MEDI-534, Cohort 1 — Participants aged 6 to less than (<) 24 months will receive MEDI-534, 10^5 median tissue culture infectious dose (TCID50) by intranasal route at Month 0, 2, and 4.
  Arms: MEDI-534, Cohort 1
Other: Placebo, Cohort 1 — Participants aged 6 to <24 months will receive placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: Placebo, Cohort 1
Biological: MEDI-534, Cohort 2 — Participants aged 6 to <24 months will receive MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: MEDI-534, Cohort 2
Other: Placebo, Cohort 2 — Participants aged 6 to <24 months will receive placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: Placebo, Cohort 2
Biological: MEDI-534, Cohort 3 — Participants aged 2 months will receive MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: MEDI-534, Cohort 3
Other: Placebo, Cohort 3 — Participants aged 2 months will receive placebo matched to MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: Placebo, Cohort 3
Biological: MEDI-534, Cohort 4 — Participants aged 2 months will receive MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: MEDI-534, Cohort 4
Other: Placebo, Cohort 4 — Participants aged 2 months will receive placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: Placebo, Cohort 4
Biological: MEDI-534, Cohort 5 — Participants aged 2 months will receive MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: MEDI-534, Cohort 5
Other: Placebo, Cohort 5 — Participants aged 2 months will receive placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
  Arms: Placebo, Cohort 5

SUMMARY:
Primary objective of this study is to describe the safety and tolerability of multiple doses of MEDI-534 in children 6 to less than (<) 24 months of age and in infants 2 months of age.

DETAILED DESCRIPTION:
This is a Phase 1/2a, randomized, double-blind, placebo-controlled, dose-escalation, multicenter study to evaluate the safety and tolerability of multiple doses of MEDI-534 at 10^5 or 10^6 median tissue culture infectious dose (TCID50) in RSV and PIV3 seronegative children 6 to <24 months of age and at dosages of 10^4, 10^5 or 10^6 TCID50 in unscreened infants 2 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female whose age on the day of randomization falls within one of the two age groups:

  6 to less than (<) 24 months (more than [>] 6 months of age and not yet reached their 2nd year birthday), Cohorts 1 and 2 2 months (+/- 4 weeks), Cohorts 3, 4, and 5
* Cohorts 1 and 2 only: Subject is seronegative to both Respiratory Syncytial Virus (RSV) and human Parainfluenza Virus Type 3 (hPIV3) at Screening
* Subject whose gestational age was greater than or equal to (>=) 36 weeks
* Subject is in general good health with normal growth (that is, body weight greater than (>) third percentile per world health organization [WHO] simplified weight-per-age field tables
* Subject's legal representative is available by telephone
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization (if applicable) obtained from the subject's legal representative
* Subject's legal representative is able to understand and comply with the requirements of the protocol as judged by the investigator
* Subject is available to complete the follow-up period 1-year after receipt of the first dose of study vaccine
* Subject's legal representative must be willing and able to bring the subject to the study site for evaluation of respiratory illness in accordance with the protocol.

Exclusion Criteria:

* Any fever (>=100.4 degrees Fahrenheit [>=38.0 degrees Celsius], regardless of route) or lower respiratory illness within 7 days prior to randomization
* Moderate or severe nasal congestion that in the investigator's opinion could interfere with intranasal delivery of study vaccine
* Acute illness (defined as the presence of moderate or severe signs and symptoms) at the time of randomization
* Any drug therapy (chronic or other) within 7 days prior to randomization or expected receipt through the protocol-specified blood collection 28 days after each study vaccine dosing, except that infrequent use of over-the-counter medications for the systemic treatment of common childhood symptoms (that is, pain relievers, decongestants or cough suppressants) are permitted according to the judgment of the investigator
* Any current or expected receipt of immunosuppressive agents including steroids (>=2 milligram per kilogram [mg/kg] per day of prednisone or its equivalent, or >=20 milligram per day [mg/day] if the subject weighs >10 kilogram [kg], given daily or on alternate days for >=14 days); children in this category should not receive study vaccine until immunosuppressive agents including corticosteroid therapy have been discontinued for >=30 days; the use of topical steroids is permitted according to the judgment of the investigator
* History of receipt of blood transfusion or expected receipt through the protocol-specified blood collection at 28 days after final study dosing
* History of receipt of immunoglobulin products or expected receipt through the protocol-specified blood collection at 28 days after final study dosing
* Receipt of any investigational drug within 60 days prior to randomization or expected receipt through 180 days after final study dosing
* Receipt of any live virus vaccine (excluding oral polio vaccine and rotavirus vaccine) within 28 days prior to randomization or expected receipt within a 28-day window around any study vaccine dose
* Receipt of any inactivated (that is, non-live) vaccine or oral polio vaccine or rotavirus vaccine within 14 days prior to randomization or expected receipt within a 14-day window around any study vaccine dose
* Known or suspected immunodeficiency, including human immunodeficiency virus (HIV) infection
* Expected to be living in the same home or enrolled in the same classroom at day care with infants <6 months within 28 days after each dose
* Living in a household with another child who is concurrently enrolled in a study of a live viral vaccine (including this study)
* Expected contact with a pregnant caregiver within 28 days after each dose
* A household contact who is immunocompromised; the subject should also avoid close contact with immunocompromised individuals for at least 28 days after any study vaccine dose
* Expected household contact within 28 days after each dose with a health care provider for immunocompromised subjects or who is a day care provider for infants under the age of 6 months
* History of allergic reaction to any component of the study vaccine
* Previous medical history, or evidence, of an intercurrent or chronic illness that, in the opinion of the investigator, may compromise the safety of the subject
* Known or suspected active or chronic hepatitis infection
* History of medical diagnosis of asthma, reactive airway disease, wheezing requiring medication, cystic fibrosis, bronchopulmonary dysplasia, chronic pulmonary disease, medically confirmed apnea, hospitalization for respiratory illness or mechanical ventilation for respiratory illness (excludes elective mechanical ventilation during surgery for subjects in Cohorts 1 and 2)
* Family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study
* Any condition that, in the opinion of the investigator, might interfere with study vaccine evaluation.

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1338 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Malkin, D.O., Study Director — MedImmune LLC
Locations (90):
- United States (47):
  - Research Site, Mobile, Alabama
  - Research Site, Bentonville, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Bell Gardens, California
  - Research Site, Downey, California
  - Research Site, Lakewood, California
  - Research Site, Long Beach, California
  - Research Site, Paramount, California
  - Research Site, San Diego, California
  - Research Site, West Covina, California
  - Research Site, Thornton, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Dalton, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Saint Paul, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, Johnson City, New York
  - Research Site, Lake Success, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, New Bern, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Gresham, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Poteet, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tomball, Texas
  - Research Site, Layton, Utah
  - Research Site, Orem, Utah
  - Research Site, St. George, Utah
  - Research Site, Midlothian, Virginia
  - Research Site, Huntington, West Virginia
- Australia (4):
  - Research Site, Garran, Australian Capital Territory
  - Research Site, Herston, Queensland
  - Research Site, North Adelaide, South Australia
  - Research Site, Subiaco, Western Australia
- Brazil (7):
  - Research Site, Passo Fundo-RS, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, Porto Alegre - RS
  - Research Site, Porto Alegre/RS
  - Research Site, Ribeirao Preto - SP
  - Research Site, Sao Paulo - SP
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Brampton, Ontario
  - Research Site, Saskatoon, Saskatchewan
- Finland (9):
  - Research Site, Helsinki
  - Research Site, Jarvenpaa
  - Research Site, Kokkola
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Tampere
  - Research Site, Turku
- Germany (3):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Mainz
- Research Site, Netanya, Israel
- South Africa (4):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Belle Ville Cape Town, Western Cape
  - Research Site, Cape Town, Western Cape
- Spain (13):
  - Research Site, Almería, Andalusia
  - Research Site, Jerez de la Frontera, Andalusia
  - Research Site, Donostia / San Sebastian, Basque Country
  - Research Site, Barcelona, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Madrid, Madrid, Communidad de
  - Research Site, Málaga, Málaga
  - Research Site, Catarroja, Valencia
  - Research Site, La Eliana, Valencia, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Esplugues de Llobregat
  - Research Site, Valencia

REFERENCES:
- [Derived] Yang CF, Wang CK, Malkin E, Schickli JH, Shambaugh C, Zuo F, Galinski MS, Dubovsky F; Study Group; Tang RS. Implication of respiratory syncytial virus (RSV) F transgene sequence heterogeneity observed in Phase 1 evaluation of MEDI-534, a live attenuated parainfluenza type 3 vectored RSV vaccine. Vaccine. 2013 Jun 10;31(26):2822-7. doi: 10.1016/j.vaccine.2013.04.006. Epub 2013 Apr 16. PMID 23602668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 720 participants were randomized in the study. An additional 618 participants were screened but not randomized in the study.
Groups:
- MEDI-534, Cohort 1: Participants aged 6 to less than (<) 24 months received MEDI-534, 10^5 median tissue culture infectious dose (TCID50) by intranasal route at Month 0, 2, and 4.
- Placebo, Cohort 1: Participants aged 6 to <24 months received placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
- MEDI-534, Cohort 2: Participants aged 6 to <24 months received MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
- Placebo, Cohort 2: Participants aged 6 to <24 months received placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
- MEDI-534, Cohort 3: Participants aged 2 months received MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
- Placebo, Cohort 3: Participants aged 2 months received placebo matched to MEDI-534, 10^4 TCID50 by intranasal route at Month 0, 2, and 4.
- MEDI-534, Cohort 4: Participants aged 2 months received MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
- Placebo, Cohort 4: Participants aged 2 months received placebo matched to MEDI-534, 10^5 TCID50 by intranasal route at Month 0, 2, and 4.
- MEDI-534, Cohort 5: Participants aged 2 months received MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
- Placebo, Cohort 5: Participants aged 2 months received placebo matched to MEDI-534, 10^6 TCID50 by intranasal route at Month 0, 2, and 4.
Period: Overall Study
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Started | 79 | 81 | 80 | 80 | 40 | 40 | 82 | 78 | 81 | 79
Treated | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
Completed | 71 | 71 | 74 | 71 | 36 | 37 | 82 | 76 | 75 | 69
Not Completed | 8 | 10 | 6 | 9 | 4 | 3 | 0 | 2 | 6 | 10
Not completed — Withdrawal by Subject | 4 | 3 | 3 | 7 | 1 | 0 | 0 | 2 | 4 | 6
Not completed — Lost to Follow-up | 3 | 6 | 3 | 2 | 3 | 3 | 0 | 0 | 2 | 3
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5 | Total
Number analyzed (Participants) | 79 | 81 | 80 | 80 | 40 | 40 | 82 | 78 | 81 | 79 | 720
Age, Customized [Number; unit: participants]
  Less than (<) 6 months | 0 | 0 | 0 | 0 | 40 | 40 | 82 | 78 | 81 | 79 | 400
  6 to <24 months | 79 | 81 | 80 | 80 | 0 | 0 | 0 | 0 | 0 | 0 | 320
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 35 | 40 | 21 | 18 | 47 | 41 | 39 | 43 | 360
  Male | 39 | 45 | 45 | 40 | 19 | 22 | 35 | 37 | 42 | 36 | 360

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Symptoms After Dose 1
Description: Solicited symptoms were predefined symptoms or events to be specifically inquired about and assessed daily during the 28-day period after vaccine administration. The solicited symptoms included fever greater than or equal to (>=) 100.4 degrees Fahrenheit (F), runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/fussiness, oropharyngeal inflammation (laryngitis), and epistaxis.
Time Frame: Within 28 days after Dose 1
Population: Dose 1 safety population included all randomized participants who received study vaccine Dose 1 and had safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants
  Any solicited symptom | 65 | 68 | 61 | 59 | 27 | 24 | 50 | 48 | 60 | 53
  Fever: 100.4 to 101.4 degrees F | 13 | 8 | 10 | 8 | 4 | 4 | 6 | 1 | 4 | 3
  Fever: 101.5 to 103.1 degrees F | 9 | 8 | 6 | 8 | 1 | 3 | 1 | 4 | 2 | 2
  Fever: 103.2 to 104.9 degrees F | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Fever: greater than (>) 104.9 degrees F | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Runny/stuffy nose | 50 | 51 | 50 | 40 | 19 | 15 | 30 | 36 | 30 | 30
  Cough | 27 | 30 | 33 | 24 | 11 | 8 | 19 | 22 | 17 | 19
  Drowsiness | 26 | 29 | 21 | 21 | 10 | 9 | 15 | 13 | 16 | 22
  Loss of appetite/decreased urine output | 22 | 26 | 21 | 21 | 7 | 7 | 9 | 6 | 12 | 12
  Irritability/fussiness | 40 | 46 | 41 | 44 | 16 | 14 | 29 | 18 | 41 | 32
  Oropharyngeal inflammation | 9 | 12 | 7 | 8 | 2 | 2 | 5 | 7 | 3 | 6
  Epistaxis | 4 | 0 | 4 | 5 | 1 | 1 | 2 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Solicited Symptoms After Dose 2
Description: Solicited symptoms were predefined symptoms or events to be specifically inquired about and assessed daily during the 28-day period after vaccine administration. The solicited symptoms included fever >=100.4 degrees F, runny/stuffy nose, cough, drowsiness, loss of appetite/decreased urine output, irritability/fussiness, oropharyngeal inflammation (laryngitis), and epistaxis.
Time Frame: Within 28 days after Dose 2
Population: Dose 2 safety population included all randomized participants who received study vaccine Dose 2 same as Dose 1 and had safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 63 | 65 | 66 | 65 | 25 | 26 | 76 | 71 | 73 | 70
participants
  Any solicited symptom | 50 | 53 | 53 | 45 | 12 | 19 | 38 | 42 | 39 | 41
  Fever: 100.4 to 101.4 degrees F | 16 | 17 | 10 | 11 | 1 | 2 | 8 | 4 | 1 | 3
  Fever: 101.5 to 103.1 degrees F | 13 | 10 | 9 | 8 | 0 | 1 | 3 | 1 | 1 | 0
  Fever: 103.2 to 104.9 degrees F | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Fever: >104.9 degrees F | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Runny/stuffy nose | 41 | 35 | 38 | 34 | 10 | 15 | 25 | 30 | 25 | 24
  Cough | 16 | 23 | 28 | 22 | 2 | 7 | 15 | 21 | 20 | 20
  Drowsiness | 20 | 13 | 15 | 15 | 5 | 4 | 11 | 7 | 7 | 10
  Loss of appetite/decreased urine output | 16 | 17 | 14 | 17 | 3 | 4 | 9 | 11 | 9 | 9
  Irritability/fussiness | 33 | 29 | 35 | 25 | 8 | 6 | 13 | 14 | 22 | 21
  Oropharyngeal inflammation | 9 | 5 | 4 | 3 | 2 | 1 | 4 | 2 | 7 | 7
  Epistaxis | 4 | 4 | 2 | 4 | 1 | 0 | 0 | 1 | 1 | 0

3. Primary Outcome: Number of Participants With Solicited Symptoms After Dose 3
Description: as for outcome 2
Time Frame: Within 28 days after Dose 3
Population: Dose 3 safety population included all randomized participants who received study vaccine Dose 3 same as previous doses and had safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 60 | 60 | 63 | 61 | 28 | 30 | 76 | 70 | 71 | 68
participants
  Any solicited symptom | 41 | 45 | 48 | 45 | 20 | 17 | 36 | 33 | 48 | 41
  Fever: 100.4 to 101.4 degrees F | 8 | 9 | 9 | 9 | 3 | 6 | 7 | 8 | 10 | 10
  Fever: 101.5 to 103.1 degrees F | 6 | 8 | 6 | 9 | 1 | 0 | 2 | 1 | 4 | 4
  Fever: 103.2 to 104.9 degrees F | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Fever: >104.9 degrees F | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Runny/stuffy nose | 36 | 35 | 35 | 28 | 16 | 15 | 24 | 21 | 32 | 31
  Cough | 22 | 14 | 20 | 17 | 10 | 10 | 14 | 15 | 25 | 23
  Drowsiness | 12 | 9 | 11 | 9 | 2 | 6 | 4 | 4 | 7 | 9
  Loss of appetite/decreased urine output | 13 | 15 | 8 | 11 | 8 | 4 | 8 | 10 | 11 | 11
  Irritability/fussiness | 23 | 25 | 29 | 28 | 11 | 8 | 11 | 11 | 20 | 14
  Oropharyngeal inflammation | 9 | 4 | 4 | 2 | 1 | 3 | 2 | 4 | 8 | 6
  Epistaxis | 2 | 1 | 2 | 4 | 0 | 2 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After Dose 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAEs) for Dose 1 are events between administration of Dose 1 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TEAEs (spontaneously reported events) after Dose 1 were reported.
Time Frame: Within 28 days after Dose 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants | 51 | 51 | 47 | 35 | 15 | 15 | 20 | 26 | 29 | 21

5. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After Dose 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-Emergent Adverse Events (TEAEs) for Dose 2 are events between administration of Dose 2 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TEAEs (spontaneously reported events) after Dose 2 were reported.
Time Frame: Within 28 days after Dose 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 63 | 65 | 66 | 65 | 25 | 26 | 76 | 71 | 73 | 70
participants | 31 | 41 | 31 | 27 | 9 | 10 | 21 | 21 | 25 | 24

6. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After Dose 3
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-Emergent Adverse Events (TEAEs) for Dose 3 are events between administration of Dose 3 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TEAEs (spontaneously reported events) after Dose 3 were reported.
Time Frame: Within 28 days after Dose 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 60 | 60 | 63 | 61 | 28 | 30 | 76 | 70 | 71 | 68
participants | 34 | 35 | 33 | 25 | 11 | 10 | 25 | 22 | 29 | 27

7. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) After Dose 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-Emergent Serious Adverse Events (TESAEs) are serious events between administration of Dose 1 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TESAEs (spontaneously reported events) after Dose 1 were reported.
Time Frame: Within 28 days after Dose 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

8. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) After Dose 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-Emergent Serious Adverse Events (TESAEs) are serious events between administration of Dose 2 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TESAEs (spontaneously reported events) after Dose 2 were reported.
Time Frame: Within 28 days after Dose 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 63 | 65 | 66 | 65 | 25 | 26 | 76 | 71 | 73 | 70
participants | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

9. Primary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) After Dose 3
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-Emergent Serious Adverse Events (TESAEs) are serious events between administration of Dose 3 and up to 28 days after the dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TESAEs (spontaneously reported events) after Dose 3 were reported.
Time Frame: Within 28 days after Dose 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 60 | 60 | 63 | 61 | 28 | 30 | 76 | 70 | 71 | 68
participants | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

10. Primary Outcome: Number of Participants With Medically-Attended Lower Respiratory Illnesses (MA-LRIs) After Dose 1
Description: An MA-LRI was a healthcare provider-confirmed diagnosis of one or more of the following events: wheezing, pneumonia, croup (laryngotracheobronchitis), rhonchi (not cleared with cough or suctioning), rales (not cleared with cough or suctioning), bronchitis, bronchiolitis, and apnea.
Time Frame: Within 28 days after Dose 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants | 2 | 2 | 4 | 4 | 0 | 0 | 1 | 0 | 0 | 2

11. Primary Outcome: Number of Participants With Medically-Attended Lower Respiratory Illnesses (MA-LRIs) After Dose 2
Description: as for outcome 10
Time Frame: Within 28 days after Dose 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 63 | 65 | 66 | 65 | 25 | 26 | 76 | 71 | 73 | 70
participants | 3 | 3 | 1 | 3 | 1 | 2 | 0 | 2 | 3 | 1

12. Primary Outcome: Number of Participants With Medically-Attended Lower Respiratory Illnesses (MA-LRIs) After Dose 3
Description: as for outcome 10
Time Frame: Within 28 days after Dose 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 60 | 60 | 63 | 61 | 28 | 30 | 76 | 70 | 71 | 68
participants | 3 | 0 | 7 | 3 | 2 | 2 | 1 | 1 | 7 | 4

13. Secondary Outcome: Number of Participants Who Shed Vaccine-Type Virus
Description: Nasal wash specimens were collected to assess vaccine virus recovery in the upper respiratory tract on 7, 12 and 28 days after each dosing.
Time Frame: 7, 12 and 28 days after Dose 1, 2 and 3
Population: Shedding population included all randomized participants who received study vaccine and had valid shedding data after the specified dose. 'N' (number of participants analyzed) = participants who were evaluable for this measure; and 'n' = participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 76 | 78 | 78 | 79 | 40 | 40 | 82 | 77 | 78 | 76
participants
  Dose 1: Day 7 (n=76,76,78,79,40,39,82,77,78,75) | 33 | 0 | 41 | 0 | 22 | 0 | 50 | 0 | 52 | 0
  Dose 1: Day 12 (n=75,78,78,78,40,40,81,76,78,76) | 21 | 0 | 14 | 0 | 16 | 0 | 29 | 0 | 22 | 0
  Dose 1: Day 28 (n=76,77,77,78,39,40,82,76,77,76) | 2 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 5 | 0
  Dose 2: Day 7 (n=62,65,65,63,25,26,75,70,72,68) | 9 | 0 | 6 | 0 | 5 | 0 | 20 | 0 | 13 | 0
  Dose 2: Day 12 (n=63,65,65,64,25,25,76,71,72,68) | 2 | 0 | 1 | 0 | 3 | 0 | 7 | 0 | 4 | 0
  Dose 2: Day 28 (n=63,65,65,65,25,26,76,71,73,68) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Day 7 (n=58,59,62,59,28,30,75,70,69,68) | 6 | 0 | 1 | 0 | 4 | 1 | 18 | 0 | 11 | 0
  Dose 3: Day 12 (n=59,60,61,61,28,29,76,70,70,68) | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 4 | 0
  Dose 3: Day 28 (n=60,60,63,61,28,30,76,70,71,68) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With a Seroresponse to Respiratory Syncytial Virus (RSV) and Human Parainfluenza Virus Type 3 (hPIV3) After Dose 3
Description: Seroresponse was defined as a >=4-fold rise from Baseline in neutralizing antibody titer, regardless of Baseline serostatus. Respiratory Syncytial Virus (RSV) and hPIV3 antibody titers were determined by using microneutralization assay and hemagglutination inhibition assay, respectively. Clopper-pearson exact confidence interval was reported.
Time Frame: Day 28 after Dose 3
Population: Immunogenicity population included all randomized participants who received study vaccine for the specified dose and had valid immunogenicity data. 'N' (number of participants analyzed) = participants evaluable for this measure; and 'n' = participants evaluable for specified virus type, for each group, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 55 | 53 | 51 | 53 | 20 | 22 | 68 | 59 | 63 | 61
percentage of participants
  RSV (n=44, 51, 50, 51, 19, 19, 68, 59, 63, 61) | 29.5 [16.8 to 45.2] | 17.6 [8.4 to 30.9] | 36.0 [22.9 to 50.8] | 25.5 [14.3 to 39.6] | 15.8 [3.4 to 39.6] | 5.3 [0.1 to 26.0] | 7.4 [2.4 to 16.3] | 3.4 [0.4 to 11.7] | 0.0 [0.0 to 5.7] | 0.0 [0.0 to 5.9]
  hPIV3 (n=55, 53, 51, 53, 20, 22, 65, 59, 57, 52) | 67.3 [53.3 to 79.3] | 7.5 [2.1 to 18.2] | 86.3 [73.7 to 94.3] | 11.3 [4.3 to 23.0] | 35.0 [15.4 to 59.2] | 4.5 [0.1 to 22.8] | 16.9 [8.8 to 28.3] | 5.1 [1.1 to 14.1] | 19.3 [10.0 to 31.9] | 5.8 [1.2 to 15.9]

15. Secondary Outcome: Genotypic Stability of Recovered Vaccine-Type Virus
Description: Nasal wash samples with vaccine-type virus were evaluated for genotypic stability, defined as the presence of the entire RSV-Fusion (RSV F) insert based on the RSV F sequence results. If the insert was absent or truncated, the recovered virus was counted as genotypically unstable. Nasal wash samples were categorized as genotypically stable, genotypically unstable or undetermined genotypic stability.
Time Frame: Within 28 days after any dose
Population: Shedding population included all randomized participants who received study vaccine and had valid shedding data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: nasal wash samples
Units Other Than Participants: nasal wash samples
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 53 | 0 | 48 | 0 | 29 | 1 | 67 | 0 | 60 | 0
Number analyzed (nasal wash samples) | 81 | 0 | 67 | 0 | 59 | 1 | 141 | 0 | 117 | 0
nasal wash samples
  Genotypically stable | 77 |  | 67 |  | 54 | 1 | 135 |  | 110 |
  Genotypically unstable | 0 |  | 0 |  | 0 | 0 | 0 |  | 0 |
  Undetermined genotypic stability | 4 |  | 0 |  | 5 | 0 | 6 |  | 7 |

16. Secondary Outcome: Number of Participants With Medically-Attended Lower Respiratory Illnesses (MA-LRIs) Through 365 Days After Randomization
Description: An MA-LRI was a healthcare provider-confirmed diagnosis of one or more of the following events: wheezing, pneumonia, croup (laryngotracheobronchitis), rhonchi (not cleared with cough or suctioning), rales (not cleared with cough or suctioning), bronchitis, bronchiolitis, and apnea. MA-LRIs occurring within 28 days post any dose and after 28 days post any dose were summarized separately.
Time Frame: Day 0 to Day 365
Population: Safety population included all randomized participants who received study vaccine and had any safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants
  Within 28 days post any dose | 8 | 5 | 12 | 10 | 3 | 4 | 2 | 3 | 10 | 7
  After 28 days post any dose | 16 | 16 | 18 | 10 | 6 | 7 | 13 | 20 | 23 | 15

17. Secondary Outcome: Number of Participants With Significant New Medical Conditions (SNMCs) Through 365 Days After Randomization
Description: An SNMC was a newly diagnosed medical condition that was of a chronic, ongoing nature and was assessed by the investigator as medically significant. Examples of SNMCs include diabetes, asthma, autoimmune disease (for example, lupus, rheumatoid arthritis), and neurological disease (for example, epilepsy, autism).
Time Frame: Day 0 to Day 365
Population: Safety population included all randomized participants who received study vaccine and had any safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1

18. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) Through 365 Days After Randomization
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-Emergent Serious Adverse Events (TESAEs) are serious events after administration of drug which were absent before treatment or that worsened relative to pretreatment state. Number of participants with unsolicited TESAEs (spontaneously reported events) within 365 days after randomization were reported.
Time Frame: Day 0 to Day 365
Population: Safety population included all randomized participants who received study vaccine and had any safety follow-up data.
Measure: Number; unit: participants
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Number analyzed (Participants) | 78 | 79 | 80 | 80 | 40 | 40 | 82 | 77 | 80 | 78
participants | 6 | 5 | 5 | 1 | 1 | 2 | 3 | 4 | 9 | 3

ADVERSE EVENTS:
Time Frame: Day 0 to Day 365
Arm/Group | MEDI-534, Cohort 1 | Placebo, Cohort 1 | MEDI-534, Cohort 2 | Placebo, Cohort 2 | MEDI-534, Cohort 3 | Placebo, Cohort 3 | MEDI-534, Cohort 4 | Placebo, Cohort 4 | MEDI-534, Cohort 5 | Placebo, Cohort 5
Serious Adverse Events (participants affected / at risk) | 6/78 | 5/79 | 5/80 | 1/80 | 1/40 | 2/40 | 3/82 | 4/77 | 9/80 | 3/78
Other Adverse Events (participants affected / at risk) | 65/78 | 66/79 | 59/80 | 55/80 | 22/40 | 27/40 | 45/82 | 42/77 | 50/80 | 44/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-534, Cohort 1 (N=78) | Placebo, Cohort 1 (N=79) | MEDI-534, Cohort 2 (N=80) | Placebo, Cohort 2 (N=80) | MEDI-534, Cohort 3 (N=40) | Placebo, Cohort 3 (N=40) | MEDI-534, Cohort 4 (N=82) | Placebo, Cohort 4 (N=77) | MEDI-534, Cohort 5 (N=80) | Placebo, Cohort 5 (N=78)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Measles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-534, Cohort 1 (N=78) | Placebo, Cohort 1 (N=79) | MEDI-534, Cohort 2 (N=80) | Placebo, Cohort 2 (N=80) | MEDI-534, Cohort 3 (N=40) | Placebo, Cohort 3 (N=40) | MEDI-534, Cohort 4 (N=82) | Placebo, Cohort 4 (N=77) | MEDI-534, Cohort 5 (N=80) | Placebo, Cohort 5 (N=78)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 6 (7) | 4 (4) | 4 (4) | 3 (4) | 4 (4) | 1 (1) | 4 (4) | 7 (8) | 2 (2) | 5 (5)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 16 (26) | 17 (23) | 17 (24) | 4 (4) | 3 (5) | 4 (5) | 2 (2) | 7 (7) | 5 (7)
Flatulence (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (7) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 21 (40) | 20 (53) | 22 (44) | 15 (39) | 1 (1) | 1 (1) | 3 (4) | 7 (8) | 3 (4) | 1 (1)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 13 (20) | 10 (12) | 11 (17) | 4 (5) | 3 (3) | 3 (3) | 3 (4) | 6 (9) | 3 (4)
Vomiting projectile (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoviral conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 6 (6) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 6 (7) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 3 (4) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 5 (6) | 5 (5) | 5 (8) | 7 (13)
Omphalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 4 (4) | 4 (4) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 11 (16) | 11 (16) | 11 (12) | 14 (15) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 2 (2)
Otitis media acute (Infections and infestations) | 7 (7) | 10 (12) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 6 (7) | 3 (3) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 4 (4) | 4 (5) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 3 (3)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (19) | 26 (31) | 22 (29) | 13 (14) | 4 (5) | 7 (7) | 15 (18) | 12 (13) | 14 (18) | 14 (17)
Viral infection (Infections and infestations) | 4 (5) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 6 (9) | 4 (4) | 9 (9) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 4 (7) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (9) | 5 (6) | 5 (7) | 1 (2) | 4 (4) | 2 (2) | 3 (3) | 6 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 6 (8) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6) | 2 (2) | 5 (6) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 5 (5) | 2 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.